CLINICAL TRIAL: NCT02673320
Title: Prospective Study for Delay in Surgical Treatment of Traumatic Cervical Central Cord Injury in Canal Stenosis
Acronym: DS3CS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC15_0040
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Acute Traumatic Cervical Central Cord Syndrom Injury
Keywords: Acute Traumatic Cervical Central Cord Syndrom Injury; Delay of Surgery; Decompressive Surgery; Canal Stenosis; Schneider Syndrom; Quality of life; Functional Outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early surgery (Experimental): Early surgery within 48 hours
  Interventions: Procedure: Early surgery within 48 hours
- Delayed surgery (Other): Delayed surgery at 15 days
  Interventions: Procedure: Delayed surgery at 15 days

INTERVENTIONS:
Procedure: Early surgery within 48 hours — After completion of the clinical and radiological diagnosis of post-traumatic spinal cord contusion on narrow spinal canal, the patient was hospitalized. After obtaining the signed consent form, the patient was included in the protocol. After anesthetic consultation determining the feasibility or not of surgery and in the absence of other vital injury or involving life-threatening, early surgery is then realised within 48 hours. The surgical technique is a conventional cervical spinal decompression surgery. Surgery by way posterior surgery, by laminectomy in case of significant spinal stenosis greater than or equal to 3 floors will be preferred. In other cases, the type of surgery will be at the discretion of the surgeon. Then, the follow-up visits are D7, M3, Y1 and Y2.
  Arms: Early surgery
Procedure: Delayed surgery at 15 days — After completion of the clinical and radiological diagnosis of post-traumatic spinal cord contusion on narrow spinal canal, the patient was hospitalized. After obtaining the signed consent form, the patient was included in the protocol. After anesthetic consultation determining the feasibility or not of surgery and in the absence of other vital injury or involving life-threatening, delayed surgery is then realised at 15 days. The surgical technique is a conventional cervical spinal decompression surgery. Surgery by way posterior surgery, by laminectomy in case of significant spinal stenosis greater than or equal to 3 floors will be preferred. In other cases, the type of surgery will be at the discretion of the surgeon. Then, the follow-up visits are D7, M3, Y1 and Y2.
  Arms: Delayed surgery

SUMMARY:
The studied pathology concerns post traumatic cervical spinal cord contusion on narrow spinal canal.

The pathophysiology remains controversial. This pathology does not enjoy consensus support. Many questions remain regarding the surgical care and its delay.

The purpose of the study was to demonstrate non-inferiority of early surgical treatment compared to the same surgery performed with a delay among patients identified as having a cervical spinal cord contusion on posttraumatic narrowed cervical canal.

In the current state of knowledge and practices, the treatment of post traumatic spinal cord contusions on narrow spinal canal spinal decompression is performed remote diagnosis. The generally accepted delay is 15 days.

The surgical technique is a conventional cervical spinal decompression surgery. The type of decompression (anterior or posterior) is dependent on the compression and therefore the clinical radiological analysis. The choice of the technique and the surgical approach are therefore left to the discretion of the surgeon.

After completion of the clinical and radiological diagnosis of post-traumatic spinal cord contusion on narrow spinal canal, the patient was hospitalized in intensive care or in the Neurosurgery Service of the University Hospital concerned.

After anesthetic consultation determining the feasibility or not of surgery and in the absence of other vital injury or involving life-threatening, early surgery within 48 hours of diagnosis is then considered (according to the assigned group).

The surgical technique is a conventional cervical spinal decompression surgery. Way posterior surgery, laminectomy for spinal stenosis significant if greater than or equal to 3 floors will be preferred. In other cases, the type of surgery will be at the discretion of the surgeon and the opinion of the Staff Neurosurgery.

The surgical procedure is identical in the two groups. Alone, the delay of the surgery varies : less than 48 hours for the first group and 15 days for the second.

During the different monitoring visits (D0 (surgery), D7, M3, Y1 and Y2), the following criteria will be assessed : the quality and quickness of the motor and sensory recovery, the early post-operative evolution and the long and medium term evolution but also disability and functional sequelaes.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman,
* Aged from 18 years old or over,
* Initial glasgow score ≥ 13,
* Initial ASIA score grade A-D,
* Scan of the cervical spine in bone windows
* Posttraumatic cervical spinal cord contusion on narrow cervical canal confirmed by MRI,
* Complete or incomplete tetraplegia on whiplash on narrow cervical canal,
* Patient's consent form (or, if appropriate, by an third party independent of the sponsor and the investigator in the case of physical disability to sign)
* Location of the stepped spinal cord injury C2 to t1,
* Affiliation to a social security system.

Exclusion Criteria:

* Nontraumatic narrow cervical canal,
* Nontraumatic not acute cervical myelopathy,
* Cervico brachial neuralgia,
* Contraindication to one of the methods studied, of a functional exploration, subject on exclusion period,
* Penetrating cervical-spinal wounds,
* Lesions threatening the vital prognosis and preventing the emergency decompression,
* Contraindications to MRI : Pacemaker or implantable defibrillator or pacemaker neurosensory, cochlear implants, ocular or cerebral ferromagnetic foreign body close to the nerve structures, metal prostheses, agitation of the patient : not cooperating or agitated patients, claustrophobic subjects, valves of neurosurgical ventriculoperitoneal shunt, dental braces,
* Pregnant women,
* Unconscious patients whose score ASIA is not feasible,
* Adults under a legal protection regime (guardianship, trusteeship, safeguard justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Score ASIA (American Spinal Injury Association) | 2 years
  Assessment of the motor skills of upper and lower limbs using the score ASIA (American Spinal Injury Association). The primary outcome measure is the Total Motor Score (Score ASIA) at 2 years : difference between the initial score ASIA at the inclusion visit and the score ASIA at 2 years. This is a functional scale divided into four assessment parameters (motor assessment, perineal assessment, functional assessment - neurological level and sensory evaluation.
  The realization of the ASIA score evaluates functional disability of a patient.

SECONDARY OUTCOMES:
Score ASIA (American Spinal Injury Association) | Day 0, Day 7, Month 3, Year 1 and Year 2
  Assessment of the motor skills of upper and lower limbs using the score ASIA. Differences between the score ASIA at the different follow-up visits (D0, D7, M3, Y1 and Y2).
Score WISCI II (Walking Index of Spinal Cord Injury) | Day 0, Day 7, Month 3, Year 1 and Year 2
  Assessment of the walking index of spinal cord injury using the WISCI II. Differences between the score WISCI II at the different follow-up visits (D0, D7, M3, Y1 and Y2).
Score SCIM III (Spinal Cord Independence Measure) | Day 0, Day 7, Month 3, Year 1 and Year 2
  Assessment of the overall functional abilities of Spinal Cord Injury using the score SCIM III (Spinal Cord Independence Measure). Differences between the score SCIM III at the different follow-up visits (D0, D7, M3, Y1 and Y2).
Score SF-36 | Day 0, Day 7, Month 3, Year 1 and Year 2
  Assessment of the quality of life using the SF-36 questionnaire. Differences between the score SF-36 at the different follow-up visits (D0, D7, M3, Y1 and Y2).
Score EVA (visual analog scale) | Day 0, Day 7, Month 3, Year 1 and Year 2
  Assessment of cervical pains using a visual analog scale. Differences between the score EVA at the different follow-up visits (D0, D7, M3, Y1 and Y2).
Score DN4 | Day 0, Day 7, Month 3, Year 1 and Year 2
  Assessment of neuropathic pains using the score DN4. Differences between the score DN4 at the different follow-up visits (D0, D7, M3, Y1 and Y2). It is a questionnaire with ten items (seven of them are issued from the patient interview and three are established by clinical examination). The DN4 questionnaire is based on the analysis of the words proposed by patients to describe their pain.
Urinary status | Day 0, Day 7, Month 3, Year 1 and Year 2
  This assessment characterizes the patient's urinary status under 4 generic items (Spontaneous micturition, reflex micturition, intermittent poll and other).
Defecation status | Day 0, Day 7, Month 3, Year 1 and Year 2
  This assessment characterizes the patient's defecation status under 4 generic items (Spontaneous defecation, reflex defecation, rectal touch and other).
Cervical spinal cord injury | Day 0, Year 1
  The data collected for each patient will be as follows : Decrease of the lesions (yes / no), disappearance of the lesions (yes / no), presence of radiological spinal cord lesion sequelae (yes / no), size of the lesion and other. The reference imaging will be the cervical spinal MRI.
Resuscitation complications | Day 0, Day 7, Month 3, Year 1 and Year 2
  Adverse events occurring during resuscitation
Decubitus complications | Day 0, Day 7, Month 3, Year 1 and Year 2
  Adverse events related to the extended position and immobility

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU d'Angers, Angers
  - CHU de Brest, Brest
  - Hospital LA TIMONE, Marseille
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No